CLINICAL TRIAL: NCT01931748
Title: Study of Non-inferiority UNCNT Versus MELSMON in Female With Menopausal Syndrome: Randomized Confirmatory Clinical Trial
Brief Title: A Randomized, Double-Blind, Parallel, Non-Inferiority, Multicenter Trial Evaluate the Efficacy and Safety of UNCNT Compared to MELSMON in Female With Menopausal Syndrome
Acronym: UNCNT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unimed Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNCNT3
Record Dates: First submitted 2013-08-21; First posted 2013-08-29 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Menopausal Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UNCNT (Experimental): 6 times/ 12 days
  Interventions: Drug: UNCNT
- MELSMON (Active Comparator): 6 times/ 12 days
  Interventions: Drug: MELSMON

INTERVENTIONS:
Drug: MELSMON
  Other Names: 6 times/ 12 days
  Arms: MELSMON
Drug: UNCNT
  Other Names: 6 times/ 12 days
  Arms: UNCNT

SUMMARY:
The Purpose of this study is to evaluate in a randomized, double-blind, Parallel, Non-inferiority, Multicenter, the efficacy and safety of UNCNT in comparison to the active comparator of MELSMON in female having menopausal syndrome. Patients will be allocated randomly to receive either UNCNT or MELSMON.

Through the injection of UNCNT to female having menopausal disorder, efficacy in the improvement of the menopausal symptoms by Kupperman index is to be evaluated and compared with MELSMON.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 40 years old
* Corresponding to one of the following criteria : Postmenopausal woman

  1. spontaneous amenorrhea for 12 month
  2. Blood serum of FSH concentration exceeds 40mlU/mL, spontaneous amenorrhea for 6month
  3. passed for at least 6 weeks of bilateral ovariectomy
  4. History of bilateral hysterectomy pasted at least 6week and blood serum of FSH more than 40mLU/ml
* Confirmed using a hot flashes recorded daily diary at visit 2: More 3-4 (times/ per day) moderate or severe flush at least a day or occurrence of more than 20 times a week to check flush
* Kupperman Index Score ≥ 15 point
* Serum Estradiol ≤ 30pg/mL
* Able to communicate to conduct the clinical trial according to the protocol
* Informed consent by oneself

Exclusion Criteria:

* Allergic to drugs or any ingredient
* Psychological menopausal disorder
* History of carcinoma such as liver cancer etc
* In the investigator's judgment, which will be unable to participate in this study

  * uncontrolled hypertensive(170/110mmHg more), severe disease (eg., of the cardiovascular, liver, kidney) or diabetic mellitus
* History of hysterectomy or bilateral ovariectomy within 6 weeks
* Patients whose blood serum AST/ALT, bilirubin and creatinine are more two times the normal maximum rate.
* Receiving hormone therapy such as estrogen, progestin or hormone of this class within a month
* Patients are participated in other clinical trials, and then receiving investigational product within 3 months.
* Usage of prohibit combination dug
* history of alcohol and drug abuse
* Washout requirement for hormone therapy such as estrogen or products involved like estrogen/progestin component ( If who has washout period of following criteria, the subject can participate in this study)

  1. hormonal vaginal formulation (ring, cream, gels, etc) ≥ 1 weeks
  2. estrogen single agent or estrogen/progestin-containing subcutaneous formulation ≥ 4 weeks
  3. Oral estrogen or progestin therapy ≥ 8 weeks
  4. Progestin intrauterine therapy ≥ 8 weeks
  5. single injection of estrogen and progestin formulation transplant ≥3 month
  6. injection of progestin or estrogen pellet method ≥ 6 month
* In woman ≥40 age, known or suspicion of breast cancer at Breast angiographic and normal pregnancy breast test within 9 month; history of breast cancer; Family history of breast cancer in one generation
* In Thickness of uterine intima ≥5mm as determined by TUVS, known or suspicion of endometrial hyperplasia or endometrial cancer by performing the endometrial biopsy
* known or suspicion of Cervical cancer in pap test ( pap smear)
* otoscleorsis
* Taking rifampicin induced liver microsome enzyme ( eg., Barbiturates, Hydantion, carbamazepine, mepeu donkey mate, John diphenyl butadiene)
* Jaundice, Dubin-Johnson syndrome or Rotor syndrome
* Vaginal bleeding for unknown reason
* Sickle cell anemia
* Severe metabolic disorder (eg., porphyria..)
* Thrombotic phlebitis, thrombosis, embolism patients, or those patients with a history
* Cerebral, coronary altery disease
* Thyroid disease, infectious disease
* Experience of using placenta drug
* Other circumstances that make the investigator expect an incomplete study participation of the patient

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Kupperman index score | baseline and 12days
  Mean difference of single clinical symptom in Kupperman index from baseline to 12days

SECONDARY OUTCOMES:
E2 | baseline and 12days
  Change in blood serum of estradiol from baseline to 12days
FSH (Folic Stimulating Hormone) | baseline and 12days
  Change in blood serum of Follicle-Stimulating Hormone from baseline to 12days.
Hot flushes | baseline and 12days
  Change in frequency and mean differences of hot flushes from baseline to 12days.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Inha Univ.Hospital,, Incheon
  - Korea University Medical center Anam Hospital, Seoul